CLINICAL TRIAL: NCT00244972
Title: Phase I Study of Tipifarnib (R115777) and Sorafenib (BAY 43-9006) in Patients With Biopsiable Advanced Cancers
Brief Title: Tipifarnib and Sorafenib Tosylate in Treating Patients With Biopsiable Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00132; NCI-2009-00132 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0363; CDR0000446569; 2005-0363 (Other: M D Anderson Cancer Center); 7156 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Sorafenib; tipifarnib

ARMS (1):
- Treatment (sorafenib tosylate, tipifarnib) (Experimental): Patients receive sorafenib tosylate PO QD or BID on days 1-28 and tipifarnib PO QD or BID on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients may be allowed to continue the treatment after the 12 courses if there is continued clinical response or disease stabilization, and patients do not have significant toxicities.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate; Drug: Tipifarnib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra

SUMMARY:
This phase I trial studies the side effects and best dose of tipifarnib when given together with sorafenib tosylate in treating patients with biopsiable cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Tipifarnib and sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity and to determine maximum tolerated dose (MTD) of tipifarnib in combination with sorafenib (sorafenib tosylate).

SECONDARY OBJECTIVES:

I. Preliminary assessment of tipifarnib and sorafenib efficacy (objective response).

II. To determine signaling pathway profiles of patients treated with tipifarnib and sorafenib who are amenable to biopsy by reverse phase protein microarray (RPPA) analysis.

OUTLINE: This is a dose-escalation study of tipifarnib.

Patients receive sorafenib tosylate orally (PO) once daily (QD) or twice daily (BID) on days 1-28 and tipifarnib PO QD or BID on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients may be allowed to continue the treatment after the 12 courses if there is continued clinical response or disease stabilization, and patients do not have significant toxicities.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had =< 4 prior chemotherapy regimens; patients must have advanced cancer that is refractory to standard therapy or for whom there is no standard therapy that increases survival by three months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (a calculated creatinine clearance [CrCL] is acceptable)
* International normalized ratio (INR)/prothrombin time (PT) =< within institutional guidelines for biopsy procedures (=< 16 seconds)
* Eligibility of patients receiving any other medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of BAY 43-9006 (sorafenib tosylate) or R115777 (tipifarnib) will be determined following review of their case by the Principal Investigator
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Tumor accessible for repeat biopsies

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any investigational agents other than BAY 43-9006 and R115777
* Patients with known brain metastases are excluded except for patients who have had treated brain metastases and are currently not taking anti-seizure medications or steroids
* Patients may not have allergies to imidazoles (e.g., clotrimazole, ketoconazole, miconazole, econazole) or a history of allergic reactions attributed to any other compound of similar chemical or biologic composition to either BAY 43-9006 or R115777
* Uncontrolled hypertension with systolic blood pressure of > 140 mmHg or diastolic pressure > 90 mmHg; however, patients with well-controlled hypertension are eligible
* Patients must not have any evidence of current history of bleeding diathesis
* Patients cannot be on therapeutic anticoagulation; prophylactic anticoagulation therapy (e.g., low-dose warfarin) of venous or arterial access devices is allowed provided that the requirements for prothrombin time (INR; international normalized ratio of prothrombin time) and partial thromboplastin time (PTT) are maintained; patients will be monitored on a weekly basis for the first (1st) cycle of treatment until the INR/PT has stabilized for 2 weeks consecutively; if patients discontinue the R115777 patients will be monitored weekly until INR/PT is stabilized for 2 weeks consecutively
* Patients may not have grade 2 or greater peripheral neuropathy
* Patients with any condition that impairs their ability to swallow pills are excluded
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs) (e.g., phenytoin, carbamazepine, phenobarbital) nor any other cytochrome P450 family 3, subfamily A, polypeptide (CYP3A4) inducer such as rifampin or St. John's wort
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a New York Heart Association (NYHA) classification > 2
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with either of these agents
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest dose level in which fewer than 2 patients experience a dose limiting toxicity as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 28 days
  Descriptive statistics and graphical analysis will be used to summarize the data. Categorical variables will be summarized in frequency tables.

SECONDARY OUTCOMES:
Clinical response evaluated using Response Evaluation Criteria In Solid Tumors criteria | Up to 4 weeks
  Descriptive statistics and graphical analysis will be used to summarize the data. For continuous variables, mean (standard deviation) or median (range) will be used to summarize outcomes.
Signaling pathway inhibition in tumor tissue by RPPA | Up to 4 weeks
  The analysis of the activated signaling pathways using Pathway Analysis (Ingenuity) will determine whether particular molecular profiles are likely to respond to tipifarnib and sorafenib.

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kurzrock R, Atkins J, Wheler J, Fu S, Naing A, Busaidy N, Hong D, Sherman S. Tumor marker and measurement fluctuations may not reflect treatment efficacy in patients with medullary thyroid carcinoma on long-term RET inhibitor therapy. Ann Oncol. 2013 Sep;24(9):2256-61. doi: 10.1093/annonc/mdt177. Epub 2013 May 14. PMID 23676418